CLINICAL TRIAL: NCT07305493
Title: The Use of Lavender (Lavandula Angustifolia) Aromatherapy Inhalation as an Anti-Anxiety Toward Pain
Brief Title: Lavender (Lavandula Angustifolia) Aromatherapy Inhalation as an Anti-Anxiety Treatment for Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitas Islam Indonesia (Other)
Responsible Party: Principal Investigator, Angga Ardhan Derryawan, MD, Principal Investigator, Universitas Islam Indonesia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 9/Ka.Kom.Et/70/KE/I/2023
Record Dates: First submitted 2025-12-12; First posted 2025-12-26 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Anxiety; Pain; Aromatherapy
Keywords: Aromatherapy; Lavandula; Anxiety; Anxiety Disorder; Pain; Mind-Body Therapies
MeSH Terms: conditions — Anxiety Disorders; Pain

STUDY DESIGN:
Intervention Model Description: This study will be plotted into two groups, consist of experimental group and controls group, participation allocation will be randomized
Who Masked: Participant, Care Provider
Masking Description: Participant will not get any information of what substances that will be the exposure or what group they are added in Care provider will received bottle A and B without any explanation what substances inside the bottle. Then the care provider will set the diffuser and diffused the substances for 30 minutes to participants
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Lavender Aromatherapy Group (Experimental): This group will be consist of 34 participants that already randomized. This group will be exposed to lavender aromatherapy
  Interventions: Combination Product: Lavender Extract Aromatherapy
- Control Group (Placebo Comparator): This control will be exposed to water diffused gas as a control to experimental group
  Interventions: Other: Placebo

INTERVENTIONS:
Combination Product: Lavender Extract Aromatherapy — This group will be exposed to diffused Lavender Extract Essential Oil Aromatherapy. Aromatherapy given to this group will be linalool concentrate (verificated with GC-MS of the essential oil) in forms of 2 mL Lavender Essential Oil from Young Living diluted in 40 mL water for 30 minutes
  Arms: Lavender Aromatherapy Group
Other: Placebo — This intervention will be just an exposure of diffused water (H2O) for 30 minutes as a control to experimental group
  Arms: Control Group

SUMMARY:
This clinical trial will assess whether aromatherapy inhalation (especially lavender extract essential oil) can be used as a complementary therapy for anxiety and pain. In this study, outcomes will be measured using the Numeric Rating Scale (NRS) for pain score and State-Trait Anxiety Inventory (STAI) questionnaire to assess state and trait anxiety scores. The two questionnaires above will be used to determine pre-post pain and anxiety scores after exposure. This study's primary research question is "Does linalool in lavender extract essential oil aromatherapy reduce anxiety in patients with pain complaints ?". With the question above, it is hypothesized that linalool can be an anti-anxiety towards pain. The product of aromatherapy will be tested in a GC-MS assay for every substance inside and proving linalool as a key substance. To prove the effect of linalool, this study will compare diffused lavender extract essential oil aromatherapy with a placebo to determine its effect as an anxiety reliever.

DETAILED DESCRIPTION:
The objective in this clinical trial is to evaluate the effect of linalool in lavender extract essential oil aromatherapy as anti-anxiety treatment for pain. The linalool inside lavender extract will be proven with GC-MS assay first. Then, after linalool has been confirmed as a key substance inside the extract, the lavender extract essential oil will be mixed with water to dilute it before it is exposed to participants in the experimental group. This study will assess anxiety and pain scale using the Numeric Rating Scale (NRS) for pain score and the State-Trait Anxiety Inventory (STAI) before exposure and 15 minutes after the exposure has been done. This complementary therapy can be an innovation in addition to conventional pain therapy, with the theory that anxiety towards pain can amplify the pain, and GABA-ergic activity in the brain can help inhibit the pain.

Study design: This study is using a Randomized Controlled Trials (RCT) with pre and post test assessment. This study will be blinding the participants and care provider.

Allocation:

* Participant will be allocated using simple randomization to the experimental or placebo group
* All the participants who agreed to the informed consent will be included and randomized to the experimental or placebo group
* Then every participant will be exposed to the intervention as scheduled personally

Group/Arm:

* Experimental Group (Lavender Aromatherapy group)
* Placebo Control Group

Intervention:

* The experimental group will use Young Living Lavender Extract Essential Oil to be diffused and exposed to participants as inhalation therapy in the experimental group. It consists 2 mL of lavender essential oil diluted in 40 mL of water (H2O). It will be exposed to participants for 30 minutes
* Placebo / Control group will be exposed to diffused water (H2O) for 30 minutes

Data Analysis Plan: The data will be analyzed using univariate analysis and bivariate analysis (Independent T-Test, Paired T-Test, Wilcoxon Test, ANOVA, and/or Mann-Whitney test)

Anticipated outcome:

* Reduction in anxiety score
* Reduction in pain score
* Low risk of allergies
* No adverse event

Risks:

* Allergies
* Adverse event

Benefits:

* Innovation in addition to pain conventional therapy as a complementary therapy
* Widely accessible
* Prices vary
* Enhances treatment and prevents reduced function or reduced quality of life

ELIGIBILITY:
Inclusion Criteria:

* Patient that complains about pain (acute or chronic) that do not have any allergic history of lavender
* Patient doesnt have any abnormalities / disease in olfactory/respiratory
* Pain are classified as moderate to severe pain (higher than 4 points in NRS)
* Patient is not in pregnant conditions

Exclusion Criteria:

* Exposure are not completed for 30 minutes due to any cause
* Consuming any pain relieving drug (such as NSAID) 1 hour before exposure or in the middle between pre and post-test period
* Any adverse event that associated to exposure or did not associated to exposure
* There is or appears to be an allergy to lavender aromatherapy ingredients.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-05-29 (Actual)

PRIMARY OUTCOMES:
Anxiety Score | Before exposure and 15 minutes after exposure has done
  This parameter measured using State Trait Anxiety Inventory (STAI) Questionnaire. This questionnaire can be used to assess state and trait anxiety. It is consist of 2 segment, state segment for current anxiety scale and trait segment for any consistent anxiety feeling scale. This questionnaire have score range between 20 (minimum) and 80 (maximum). It is classified as mild anxiety for 20-39 points, moderate anxiety for 40-59 points, and severe anxiety for 60-80 points. This questionnaire has been tested for its validity by McDowell in 2006 with interval value 0,88. For its reliability, it has been tested by McDowell too in 2006 with alpha for S part 0,93 and T part 0,91

SECONDARY OUTCOMES:
Pain Scale | Before exposure and 15 minutes after exposure has done
  This parameter measured with NRS questionnaire for assessing pre-post exposure pain scale changes. This questionnaire will have score range between 0-10 points. 0 point stands for no pain, 1-3 points will stands for mild pain, 4-6 for moderate pain, and 7-10 stands for severe pain

CONTACTS AND LOCATIONS:
Overall Officials: Angga A Derryawan, MD, Principal Investigator — Universitas Islam Indonesia
Locations (1):
- Ludira Husada Hospital, Yogyakarta, D.I.Yogyakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that will be shared will be raw data of anxiety and pain score. If requested, participant demographic data will be shared in limited information due to privacy
Supporting Information: Study Protocol, ICF
Time Frame: Supporting information will be available until end of December 2027 (4 years after the study has completed)
Access Criteria: Anyone who studying / researching and needed raw data can contact this study principal investigator to access this study raw data